CLINICAL TRIAL: NCT01129726
Title: Fiberoptic Intubation and Transillumination-guided Fiberoptic Intubation：Time and Success Rate in Untrained Medical Personnel
Brief Title: Fiberoptic Intubation and Transillumination-guided Fiberoptic Intubation：Success Rate and Time in Untrained Medical Personnel
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Second Military Medical University (Other)
Responsible Party: Principal Investigator, Yang Tao, Department of Anesthesiology and Cirtical Care Medicine, Changhai Hospital, Second Military Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: 20100002; Light Guided (Other: SMMU)
Record Dates: First submitted 2010-05-18; First posted 2010-05-25 (Estimated); Last update posted 2012-02-17 (Estimated); Status verified 2012-02

CONDITIONS: Transillumination-guided Fiberoptic Intubation Intubation
Keywords: Transillumination-guided; Fiberoptic Intubation; time; success rate; intubation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intubation (Experimental): Transillumination-guided Fiberoptic Intubation
  Interventions: Device: Transillumination-guided Fiberoptic Intubation

INTERVENTIONS:
Device: Transillumination-guided Fiberoptic Intubation — Light guided, Non-invasive
  Other Names: Light guided Bronchoscopic Intubation Technique

SUMMARY:
Fiberoptic Intubation is the preferred technique to difficult airway. However, when performed by untrained anesthesiologists, bronchoscopic intubation has a high rate of failure. We want to know if the Transillumination-guided Fiberoptic Intubation technique can improves the success rate and time for tracheal intubation performed by inexperienced anesthesiologists; whether this technique improves the success rate and for normal intubations when performed by inexperienced anesthesiologists as well is unknown. Therefore, the authors compared the success rate and time of Fiberoptic Intubation versus the Transillumination-guided Fiberoptic Intubation performed by anesthesiologists inexperienced in Fiberoptic Intubation.

ELIGIBILITY:
Inclusion Criteria:

* general anesthesia
* ASA I~II
* Mallampati Score grade I~II
* thyromental distance ≥6cm
* mouth-open ≥3cm
* body mass index (BMI) ≤30kg/m2

Exclusion Criteria:

* neck and maxillofacial surgeries
* potential risks for regurgitation and pulmonary aspiration
* in pregnancy

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2010-05; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
time to intubation | Within 3 month

SECONDARY OUTCOMES:
success rate and postoperative side effect | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: XiaoMing Deng, Ph.D., Study Chair — Second Military Medical University
Locations (2):
- China (2):
  - Changhai Hospital Affiliated to Second Military Medical University, Shanghai, Shanghai Municipality
  - Changhai Hospital affiliated to Second Military Medical University, Shanghai